CLINICAL TRIAL: NCT03249545
Title: Late Effect of Ablation on Premature Ventricular Complex Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Principal Investigator, Fırat Özcan, MD,Associate Profesor, Yuksek Ihtisas Hospital
Other Study IDs: ozcan02
Record Dates: First submitted 2017-08-06; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Premature Ventricular Complex; Electrophysiology; Ablation
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Premature Ventricular Complex (PVC) ablation is performed in certain indications. Generally acutely abolition of PVC at the time of ablation accepted as successful ablation. However in some patients this effect occurs lately. In this study investigators sought late effect of ablation

DETAILED DESCRIPTION:
On tissue level ablation lesion deepens and enlarges by time following the procedure. Based on this, investigators aimed to seek patients who has no acute success but late success. This phenomenon occurs in some patients. Investigators investigate the characteristics of those patients on both procedural and clinical aspects. Investigators enroll patients applied during prespecified dates

ELIGIBILITY:
Inclusion Criteria:

Patients who had both of the criteria below

* Presence of premature ventricular complex requiring ablation
* Successfully abolition of premature ventricular complex hours after the procedure

Exclusion Criteria:

Patients who had either of below mentioned criteria

* Abolition of premature ventricular complex during the procedure
* Unsuccessful procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals having premature complexes and matching ablation indications are included and selection will be based on above mentioned criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Success | 3 months
  Continuation of ablation on the long term

CONTACTS AND LOCATIONS:
Locations (1):
- Turkiye Yuksek Ihtisas Training and Research Hospital, Ankara, Turkey (Türkiye)